CLINICAL TRIAL: NCT01488318
Title: Phase II Trial of Cetuximab and Dasatinib in Patients With Cetuximab-resistant, Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck and Low Serum IL-6
Brief Title: Cetuximab and Dasatinib in Recurrent Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI leaving the institution
Sponsor: Julie E. Bauman, MD, MPH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Julie E. Bauman, MD, MPH, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-034; CA180264 (Other: BMS)
Record Dates: First submitted 2011-11-30; First posted 2011-12-08 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Squamous Cell Carcinoma Of The Head And Neck
Keywords: Cetuximab; Dasatinib; Squamous Cell; Head and Neck; After Cetuximab Containing Chemoradiotherapy; Recurrent; Metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — Cetuximab; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CETUXIMAB AND DASATINIB (Experimental): Cetuximab on a standard weekly schedule (see Section 6.2). Group 1 (subjects more than 2 weeks post last dose of Cetuximab): Loading dose of 400 mg/m2 on cycle 1, day 1 then 250 mg/m2 IV weekly.
  Group 2 (subjects last Cetuximab treatment within 2 weeks): Cycle 1 will start at a dose of 250 mg/m2 Dasatinib 150 mg once daily without interruption. On the FIRST cycle (1 cycle is 3 weeks) dasatinib will start 3 days after the cetuximab loading dose (i.e. cycle 1, day 4) to avoid headache as shown on the previous phase I trial.
  Treatment will continue until progression.
  Interventions: Drug: Cetuximab; Drug: Dasatinib

INTERVENTIONS:
Drug: Cetuximab — Cetuximab 250 mg/m2 IV weekly after loading dose 400 mg/m2 on cycle 1, day 1
  Other Names: Erbitux
Drug: Dasatinib — Dasatinib 150 mg po

SUMMARY:
This is a single-arm, non-masked, open-label, Phase II study of cetuximab + dasatinib in recurrent Squamous Cell Carcinoma of The Head and Neck (SCCHN) that has recurred after cetuximab-containing therapy (please see attached schema).

The primary endpoint 12-week PFS.

DETAILED DESCRIPTION:
Patients must have recurrent SCCHN and may have received any number of prior palliative systemic therapies for recurrent disease (without cetuximab or othr EGFR inhibitor). One prior curative regimen (induction, primary or postoperative chemoradiotherapy) should have been given AND all patients should have been exposed to cetuximab as part of prior potentially curative treatment.Those who have received a prior Src kinase inhibitor or EGFR inhibitor other than cetuximab are not eligible.

Patients will be tested for serum IL-6. If IL-6 is detectable, the patient will be ineligible. If IL-6 is not detected, the patient will be eligible for the study. Subjects more than 2 weeks post last dose of Cetuximab will receive an initial loading dose 400 mg/m2 on cycle 1, day 1. Subjects who have received Cetuximab within 2 weeks of starting study will start Cycle 1 with dose of 250 mg/m2. Dasatinib will start 3 days after initial cetuximab study dose on cycle 1 (i.e cycle 1, day 4), and continue without interruption.

ELIGIBILITY:
Inclusion:

* Patients must have metastatic and/or recurrent SCCHN that has been previously treated with cetuximab.
* Undetectable baseline serum IL-6 NOTE : This eligibility criterion applies only to patients enrolling to the second, biomarker-enrichment stage of the trial.
* Measurable disease per RECIST 1.1.
* Unlimited prior treatment with radiation or chemoradiotherapy
* Any number of prior regimens for recurrent or metastatic SCCHN (i.e. palliative treatment) including cetuximab or other EGFR inhibitor
* Age >18 years
* ECOG performance status <2 (Karnofsky >60%, see Appendix A).
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  1. absolute neutrophil count >1,200/µL
  2. platelets >100,000/µL
  3. total bilirubin within normal institutional limits
  4. AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
  5. Creatinine up to 1.5 X normal institutional limits
* Ability to understand and the willingness to sign a written informed Consent document.
* Patients should not be taking concomitant medication that are CYP3A4 inducers or potent inhibitors and should try to avoid taking proton pump inhibitors and H2 antagonists during rest of treatment period. The above medications will be continued only if medically necessary and their use will be noted.
* Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. All WOCBP MUST have a negative pregnancy test prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study. In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.

Exclusion:

* Patients who have not recovered from adverse events due to prior agents. A minimum interval of 3 weeks should have elapsed from prior chemotherapy other than cetuximab. A minimum of 12 weeks should have elapsed from prior definitive radiotherapy, and a minimum of 1 week should have elapsed from prior palliative radiotherapy.
* Patients may not have received an investigational agent within 4 weeks of starting this trial.
* Patients with untreated brain metastases should be excluded from this clinical trial.
* History of allergic reactions to monoclonal antibodies.
* Inability to swallow oral medications (unless patients use a feeding tube in which case they are eligible).
* Uncontrolled angina or uncontrolled hypertension or any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec) on the Bazett's correction.
* Diagnosed or suspected congenital long QT syndrome.
* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including: quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
* Any other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bauman, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stabile LP, Egloff AM, Gibson MK, Gooding WE, Ohr J, Zhou P, Rothenberger NJ, Wang L, Geiger JL, Flaherty JT, Grandis JR, Bauman JE. IL6 is associated with response to dasatinib and cetuximab: Phase II clinical trial with mechanistic correlatives in cetuximab-resistant head and neck cancer. Oral Oncol. 2017 Jun;69:38-45. doi: 10.1016/j.oraloncology.2017.03.011. Epub 2017 Apr 9. PMID 28559019
- [Derived] Gross ND, Bauman JE, Gooding WE, Denq W, Thomas SM, Wang L, Chiosea S, Hood BL, Flint MS, Sun M, Conrads TP, Ferris RL, Johnson JT, Kim S, Argiris A, Wirth L, Nikiforova MN, Siegfried JM, Grandis JR. Erlotinib, erlotinib-sulindac versus placebo: a randomized, double-blind, placebo-controlled window trial in operable head and neck cancer. Clin Cancer Res. 2014 Jun 15;20(12):3289-98. doi: 10.1158/1078-0432.CCR-13-3360. Epub 2014 Apr 11. PMID 24727329

RESULTS

PARTICIPANT FLOW:
Groups:
- CETUXIMAB + DASATINIB: Cetuximab dosed at 250 mg/m^2/week and Dasatinib dosed at 150 mg daily
Period: Overall Study
Arm/Group | CETUXIMAB + DASATINIB
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CETUXIMAB + DASATINIB
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 62 [51.7 to 72.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Number of patients experiencing a Complete Response (CR) + Partial Response (PR) to study treatment / Total number of evaluable patients, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 36 months
Population: Patients that received Cetuximab dosed at 250 mg/m^2/week and Dasatinib 150 mg daily who were evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | CETUXIMAB + DASATINIB
Number analyzed (Participants) | 13
percentage of participants | 0

2. Primary Outcome: Response to Treatment
Description: Response of evaluable patients to treatment, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 36 months
Population: Patients that received Cetuximab dosed at 250 mg/m^2/week and Dasatinib 150 mg daily who were evaluable for response.
Measure: Number; unit: participants
Arm/Group | CETUXIMAB + DASATINIB
Number analyzed (Participants) | 13
participants
  Patients experiencing Stable Disease (SD) | 5
  Patients experiencing Progressive Disease (PD) | 8

3. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 36 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CETUXIMAB + DASATINIB
Number analyzed (Participants) | 14
months | 1.7 [1.4 to 3.9]

4. Secondary Outcome: Overall Survival (OS)
Description: From date of entry into the study until the date of death from any cause, assessed up to 60 months.
Time Frame: Up to 60 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CETUXIMAB + DASATINIB
Number analyzed (Participants) | 14
months | 5.1 [4.2 to 11.5]

ADVERSE EVENTS:
Arm/Group | CETUXIMAB + DASATINIB
All-Cause Mortality (participants affected / at risk) | 8/14
Serious Adverse Events (participants affected / at risk) | 8/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CETUXIMAB + DASATINIB (N=14)
Edema face (General disorders) | 1
Edema limbs (General disorders) | 1
Fever (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Injury to carotid artery (Injury, poisoning and procedural complications) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CETUXIMAB + DASATINIB (N=14)
Leukocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Facial pain (General disorders) | 1
Flu like symptoms (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Weight loss (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Movements involuntary (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Lymphedema (Vascular disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Aspartate aminotransferase increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Platelet count decreased (Investigations) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Fatigue (General disorders) | 6
Pain (General disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
Lymphocyte count decreased (Investigations) | 8
Anemia (Blood and lymphatic system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes